CLINICAL TRIAL: NCT04236362
Title: A Phase Ib, Single Arm, Open-label Study of TQB2450 Combined With Anlotinib in Subjects With Relapsed / Refractory Gynecological Cancer
Brief Title: A Study of TQB2450 Combined With Anlotinib in Subjects With Gynecological Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-10
Record Dates: First submitted 2020-01-18; First posted 2020-01-22 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Gynecological Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450+Anlotinib (Experimental): TQB2450 1200 mg IV on Day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor

SUMMARY:
This is a single-arm, open-label, phase Ib clinical trial to evaluate the efficacy and safety of TQB2450 combined with anlotinib in subjects with gynecological cancer, including 34 ovarian cancer，34 endometrial cancer，22 cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Understood and signed an informed consent form;
2. 18 years and older, male or female, Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, life expectancy ≥ 3 months;
3. Histologically confirmed, unresectable recurrent/metastatic advanced gynecologic cancer, including ovarian, endometrial, and cervical cancer;
4. Subjects have received at least 1 line platinum-containing chemotherapy (minimum of 4 cycles of platinum-containing treatment) after tumor reduction, and meet any of the following：Platinum-resistant or refractory patients, including patients who have progressed or relapsed during previous platinum-containing chemotherapy regimens or within 6 months after the end of platinum-containing chemotherapy;
5. At least one measurable lesion according to the RECIST 1.1;
6. The main organs function are normally;
7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

1. Has other non-epithelial ovarian tumors or borderline ovarian epithelial tumors;
2. Other malignant tumors that have appeared or are currently present within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors;
3. Has previously received immune drugs such as PD-1 / PD-L1, CTLA-4 or other tyrosine kinase inhibitors such as anlotinib hydrochloride;
4. Has received bevacizumab within 28 days before the first dose;
5. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks;
6. Expect to use any active vaccine against infectious diseases (such as influenza vaccine, chickenpox vaccine, etc.) within 28 days before the first dose or during the study period;
7. Patients diagnosed with immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose> 10mg / day prednisone or other effective hormones) and continue to use it within 2 weeks before the first dose;
8. Active autoimmune diseases that require systemic treatment have occurred within 2 years before the first dose;
9. Subjects known to be allergic to the study drug or any of its excipients or have experienced a severe allergic reaction to other monoclonal antibodies;
10. Has uncontrollable symptoms of brain metastases, spinal cord compression, cancerous meningitis;
11. Has any bleeding or bleeding event ≥ CTC AE Grade 3 or unhealed wounds, ulcers or fractures within 4 weeks before the first dose;
12. Has clinically significant thyroid dysfunction before the first dose;
13. Has multiple factors affecting oral medication;
14. Has any severe acute complications before the first dose;
15. Has participated in other anti-tumor intervention clinical trials within 4 weeks before the first medication;
16. According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases including mental disorders need to be treated together, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR)

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  Time from tumor first assessment to CR or PR to first assessment to PD (Progressive Disease) or death from any cause
Disease control rate（DCR） | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Overall Survival (OS) | up to 120 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei

REFERENCES:
- [Derived] Lan CY, Zhao J, Yang F, Xiong Y, Li R, Huang Y, Wang J, Liu C, Bi XH, Jin HH, Meng J, Zhao WH, Zhang L, Wang YF, Zheng M, Huang X. Anlotinib combined with TQB2450 in patients with platinum-resistant or -refractory ovarian cancer: A multi-center, single-arm, phase 1b trial. Cell Rep Med. 2022 Jul 19;3(7):100689. doi: 10.1016/j.xcrm.2022.100689. PMID 35858589